CLINICAL TRIAL: NCT03437408
Title: Influence of Ventricular Pacing on Automated Ventricular Substrate Mapping and Relationship Between Ablation Index and Impedance Drop in the Human Ventricle
Brief Title: Late Potentials and Ablation Index in Ventricular Tachycardia Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RHM CAR0538
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Catheter Ablation; Late Potential; Ablation Index; Pacing
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Ventricular Substrate maps in patients undergoing ablation for VT - maps collected with automated tagging in different pacing modalities. Validation of collected substrate. Collection of impedance and ablation index data during ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mapping and ablation (Experimental): Automated Substrate maps with different pacing modes. Validation of collected substrate. Data collection during ablation
  Interventions: Device: Mapping and ablation

INTERVENTIONS:
Device: Mapping and ablation — High density substrate map. Data collection during ablation

SUMMARY:
There is an increasing evidence regarding the efficacy of a substrate-based ablation approach to ventricular tachycardia (VT). This approach involves identifying regions of scar and also areas displaying late potentials and fractionated activity. Automated mapping systems are now available which may be able to generate high density maps displaying regions containing both late potentials and ventricular scar. Such an automated approach has not been validated. Furthermore, most patients presenting for VT ablation have pacing devices in situ. It is not known how the pacing modality affect the substrate maps generated for these procedures. Once an area felt to be important to ablate has been identified, the next key step is to perform effective ablation. An algorithm has now been made available (Ablation index - Biosense Webster Inc.,) which in preclinical studies is an effective predictor of radiofrequency lesion depth. This algorithm has been studied extensively in the atrium but not in the ventricle. This study would also seek to collect ablation index data during ablation to assess the algorithm during ventricular ablation.

DETAILED DESCRIPTION:
The study would propose to use the Carto3 mapping system with the Confidense automated tagging module (Biosense Webster Inc.,) and a high density mapping catheter to generate substrate maps of the ventricle, with maps generated with varying pacing modes. A SmartTouch catheter (Biosense Webster Inc.,) would then be used for ablation with data collected during each ablation.

The study hypotheses are:

* High density automated mapping systems can be used to generate accurate ventricular substrate maps.
* There will be a significant change in the late potential maps based on the presence and type of ventricular pacing.
* The relationship between impedance drop and ablation index during ablation will be stronger than FTI and will allow formulation of an upper limit for clinical ventricular ablation.
* The relationship between FTI and AI with impedance drop will be stronger than with electrogram attenuation.

Protocol:

15 patients, listed on clinical grounds for a left ventricular VT ablation in the context of structural heart disease (including redo ablation) would be recruited for the trial. All patients would need to have a pacing device in situ and have underlying sensed ventricular rhythm (with or without atrial pacing), or in the absence of a sensed ventricular rhythm, a biventricular pacing device. As part of their clinical work-up for the procedure, patients will have cardiac MRI scans wherever possible.

All procedures would be undertaken with Carto3, using a PentaRay catheter for mapping in concert with the Confidense module, and a SmartTouch or SmartTouch SF catheter for ablation (Biosense Webster).

Procedures would be conducted under moderate ('conscious') sedation or general anaesthetic.

Mapping Phase Mapping would be performed antegrade, retrograde or a combination of both. The first map taken would be without ventricular pacing using the PentaRay catheter and Confidense. Confidense maps would be displayed showing bipolar voltage and late potentials in Carto3. The aim would be for maximal coverage of the ventricle. A remap would then be undertaken with pacing from the patient's right ventricular pacing lead. In patients with an additional left ventricular lead, maps would also be made with left ventricular only and biventricular pacing. In those patient without underlying ventricular sensed rhythm, maps would be taken with right ventricular only, left ventricular only and biventricular pacing.

The automatically collected maps would then be validated. The PentaRay would be moved over to 2 areas where there is agreement between the maps over the presence of late potentials and, while the PentaRay was kept in the same place, manual points would be taken with one pacing mode and then with the pacing mode changed. This would also be repeated for 2 areas where there is disagreement over the presence of late potentials. This process would also be repeated for areas identified as showing scar. All points would be taken with respiratory gating. Off line, the areas identified as showing abnormal signal - either scar or late potentials - would be manually checked to ensure the system has correctly identified them.

Ablation Phase Ablation would be undertaken using a Smart Touch Surround Flow Catheter (Biosense Webster). Ablation power would be restricted to 40-50W based on the operator's choice. Steerable sheath usage would be encouraged but not mandatory. Each radiofrequency application would be delivered with the catheter stable prior to the ablation. A mapping point would be taken with the catheter stable, and then a static ablation would be delivered and an ablation point manually taken. Following cessation of ablation, a further mapping point would be taken. All points would be respiratory gated. Ablations would be non-overlapping. If there was displacement of the catheter during the ablation, this ablation would be removed from the impedance analysis.

Quantitative comparisons Mapping Study The percentage of the maps showing scar and late potentials would be quantitatively analysed by exporting the data from Carto3. As comparisons would be made between pacing modes, each patient would act as their own control. Based on prior work, bipolar scar would be defined as <0.5mv for dense scar and 0.5-1.5mV for low voltage areas12, while unipolar scar would be <5mV. The characteristic of the late potentials - specifically how late they were compared to the QRS and their size would be compared quantitatively for electrograms taken manually at the same location with the PentaRay. Quantitative analyses of the data exported from Carto 3 would be conducted using novel algorithms programmed in Matlab (Mathworks, Natick, MA, USA).

Ablation Study The Carto3 data export would be utilized to obtain the impedance, contact force, temperature and location data and electrogram data (pre- and post-ablation) for each ablation. These data would then be analysed using custom Matlab scripts to undertake an incremental AI and FTI based analysis of the impedance drop during ablation. The curves would then be analyzed with the target of quantitatively describing the relationships with impedance drop and if possible providing the plateau points in the curve to generate an upper limit for ablation.

Value of Results This study would assess automated electrogram collection as a valid methodology for rapidly generating ventricular substrate maps. This will help to shorten procedure times for VT ablation by guiding the physician to the areas of interest more rapidly. At present, it is unknown how the pacing mode affects substrate maps in the ventricle and consequently the mode in which to leave pacing. The study will help to guide us to maximise the appropriate identification of the VT substrate by picking the correct pacing mode for the procedure.

The study would validate the use of ablation index for clinical ventricular ablation as well as aiming to provide guidance as to how to use this for maximal safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular Tachycardia; scheduled for ablation on clinical grounds; able/willing to consent to procedure/research protocol; no contraindication to clinical ablation; ≥18 years old

Exclusion Criteria:

* Unable/unwilling to consent; contraindication to clinical ablation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Areas with ventricular tachycardia substrate | Through study completion, an average of 1 year
  Quantification of late potential area and scar area with comparison between pacing modalities

SECONDARY OUTCOMES:
Relationship between ablation index and impedance drop | Through study completion, an average of 1 year
  Quantification of the relationship between ablation index and impedance drop during ablation.
Relationship between Force Time Integral and impedance drop | Through study completion, an average of 1 year
  Quantification of the relationship between Force Time Integral and impedance drop during ablation.
Relationship between electrogram attenuation and impedance drop | Through study completion, an average of 1 year
  Quantification of the relationship between electrogram attenuation and impedance drop during ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Waqas Ullah, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Southampton General Hospital, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Derived] Bates AP, Paisey J, Yue A, Banks P, Roberts PR, Ullah W. Radiofrequency Ablation of the Diseased Human Left Ventricle: Biophysical and Electrogram-Based Analysis. JACC Clin Electrophysiol. 2023 Mar;9(3):330-340. doi: 10.1016/j.jacep.2022.10.001. Epub 2022 Oct 10. PMID 36371330